CLINICAL TRIAL: NCT02967016
Title: A Pilot Study: To Compare Physical Activity After a Normal Spontaneous or Cesarean Delivery by Use of a Actigraph GT3X
Brief Title: Physical Activity After a Normal Spontaneous or Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: George Washington University (Other)
Responsible Party: Principal Investigator, Dongchen Li, MD, Assistant Professor Director of Obstetric Anesthesia Department of Anesthesiology, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20160001283
Record Dates: First submitted 2016-10-28; First posted 2016-11-17 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Postpartum Disorder
MeSH Terms: conditions — Puerperal Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal spontaneous vaginal delivery (Experimental): Both groups will be asked to wear a fitness tracker (Actigraph GT3X+).
  Interventions: Behavioral: Actigraph
- Cesarean Delivery (Experimental): Both groups will be asked to wear a fitness tracker (Actigraph GT3X+).
  Interventions: Behavioral: Actigraph

INTERVENTIONS:
Behavioral: Actigraph — following delivery a ActiGraph will be offered to patients to track their steps

SUMMARY:
To the best of the investigators knowledge the average level of physical activity (PA) of parturients recovering from a cesarean delivery or after a normal spontaneous vaginal delivery (NSVD) remains unknown. Taking in consideration that parturients are in a hypercoagulable state and that obstetric venous thromboembolism (VT) is one of the most common causes of maternal morbidity and mortality, ambulation is of utmost importance to anesthesiologists as well as obstetricians. In order to promote mobility, first the investigators need to learn the average parturients level of physical activity in the immediate post-partum period and up to 48 hours after delivery. This information may help us promote mobility in the immediate postpartum period, particularly for those that underwent a cesarean delivery since they are at higher risk of VT.

DETAILED DESCRIPTION:
Cesarean delivery is the most common surgery performed in the United States. Despite this fact, there is a paucity of literature looking into the implementation of enhanced recovery after surgery (ERAS) for patients undergoing this type of surgery. ERAS protocols have shown to improve recovery from surgery, decreasing complication and hospital length of stay. The pathway for enhanced recovery targets improving 3 factors that have been associated with increased hospital length of stay and complications. These factors are pain, immobilization and postoperative ileus. These factors, many times are inter-related. A patient in pain would tend not to ambulate as this may exacerbate the pain and discomfort. In order to alleviate pain, the patient would most likely receive an opioid for pain management and these medications are known to have undesirable side effects such as nausea, vomiting, sedation, respiratory depression, constipation and urinary retention. All of these adverse effects (AEs) may lead to complications or increased hospital length of stay.

To the best of the investigators knowledge the average level of physical activity (PA) of parturients recovering from a cesarean delivery or after a normal spontaneous vaginal delivery (NSVD) remains unknown. Taking in consideration that parturients are in a hypercoagulable state and that obstetric venous thromboembolism (VT) is one of the most common causes of maternal morbidity and mortality, ambulation is of utmost importance to anesthesiologists as well as obstetricians. In order to promote mobility, first we need to learn the average parturients level of physical acuity in the immediate post-partum period and up to 48 hours after delivery. This information may help us promote mobility in the immediate postpartum period, particularly for those that underwent a cesarean delivery since they are at higher risk of VT.

Given the lack of knowledge regarding the physical activity level of parturients in the postpartum period, the investigators have designed a pilot study to objectively measure their PA. Patients having a normal spontaneous vaginal delivery will serve as our control group. These patients are going through the same physiologic changes that their counterparts (CD patients) are going through, the only difference being the stress of surgery in the CD group.The use of Fitness trackers (i.e Fitbit(R), Actigraph GT3X +) has been used to measure and promote physical activity in a cardiac rehabilitation population, as well as in parturients self-identified as inactive. The investigators intend to use the Actigraph GT3X+ to measure the level of physical activity of 50 parturients (25 NSVD and 25 post CD). The information obtained, will help us tailor the anesthetic/analgesic management of parturients in such a way that promotes early ambulation and recovery. The investigators estimate that we need approximately a total of 50 patients, 25 per group to assess if there is a difference in the level of PA between parturients after a NSVD or CD. We will aim to recruit 60 patients 30 per group to account for missing data, protocol violations, equipment malfunction or patients drop outs.This will be a pilot, prospective study aimed at measuring the physical activity (PA) of American Society of Anesthesiologists (ASA) Classification I and II women aged 18 years and older, after a normal spontaneous vaginal (NSVD) or cesarean delivery (CD). Subjects will be ASA I and II women aged 18 years and older, knowing to have had either a NSVD or CD (under neuraxial anesthesia). After delivery, and assuring that mother and baby are stable, patients will be approached by a member of the study team to discuss the study and obtain informed consent. After obtaining informed consent, patients will be divided into Two (2) groups depending on the mode of delivery. Group 1 will be NSVD and group 2 will be CD patients. Patients will be provided with a fitbit- based Actigraph GT3X + hardware, 3 hours after delivery. Patients will be evaluated every 12 hours after delivery for a period of 48 hours. During these evaluation points, pain (visual analogue scores), factors affecting mobility, and level of satisfaction with their analgesia will be assessed. After 48 hours the Actigraph GT3X + will be interrogated and objective data, such as mean daily steps, will be obtained using the aforementioned software.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-45 years old giving birth after receiving a neuraxial analgesia/anesthesia technique. American Society of Anesthesiologists classification 1-2.

Exclusion Criteria:

* History of chronic pain
* Recent use of opioids (other than postpartum)
* Emergency case requiring general anesthesia (GA) or conversion to GA
* BMI > 45
* Need to perform more extensive surgery (i.e Hysterectomy) Need for the neonate to be admitted to NICU (This will prompt mothers to walk more frequently, and longer distances to visit the baby)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Gonzalez-Fiol, MD, Study Director — Yale New Haven Hospital
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - University Hospital, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Spontaneous Vaginal Delivery | Cesarean Delivery
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cesarean Delivery: Patients delivered via cesarean section
- Vaginal Delivery: Patients delivery via cesarean delivery
- Total: Total of all reporting groups
Arm/Group | Cesarean Delivery | Vaginal Delivery | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (5.9) | 28.3 (6.0) | 30.0 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 10 | 14 | 24
  White | 10 | 9 | 19
  Asian | 0 | 1 | 1
  Other | 4 | 1 | 5
  Not available | 1 | 0 | 1
Body Mass index [Mean (Standard Deviation); unit: Kg/m2] | 32 (6.3) | 31.4 (6.0) | 31.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Steps
Description: This will be measured in the numbers of steps registered by the accelerometer
Time Frame: from 6 hours the after delivery until discharge or 48 hours whatever happens first
Population: steps
Measure: Mean (Standard Deviation); unit: Steps
Arm/Group | Cesarean Delivery | Vaginal Delivery
Number analyzed (Participants) | 25 | 25
Steps
  6 | 968 (920) | 1771 (660)
  12 | 1652 (1206) | 3165 (1266)
  24 | 3421 (2314) | 5911 (2162)
  36 | 4919 (3678) | 8841 (3113)
  48 | 6306 (5835) | 9813 (3916)
Statistical Analysis 1: Comparison: Cesarean Delivery vs Vaginal Delivery; Cumulative Steps 6 h; Test type: Other; p = 0.002, Kruskal-Wallis
Statistical Analysis 2: Comparison: Cesarean Delivery vs Vaginal Delivery; Cumulative steps 12 h; Test type: Other; p = .0002, Kruskal-Wallis
Statistical Analysis 3: Comparison: Cesarean Delivery vs Vaginal Delivery; Cumulative steps 24 h; Test type: Other; p = .0006, Kruskal-Wallis
Statistical Analysis 4: Comparison: Cesarean Delivery vs Vaginal Delivery; Cumulative steps 36 h; Test type: Other; p = 0.0006, Kruskal-Wallis
Statistical Analysis 5: Comparison: Cesarean Delivery vs Vaginal Delivery; Cumulative steps 48 h; Test type: Other; p = 0.03, Kruskal-Wallis

2. Secondary Outcome: Pain Score at Rest
Description: This outcome will be measured using a visual analogue score (VAS). Patient will mark their pain on a 0-100 mm line with 0 been no pain and 100 mm worst pain.
Time Frame: 6 hours following delivery until 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Cesarean Delivery | Vaginal Delivery
Number analyzed (Participants) | 25 | 25
score on a scale (0-100)
  6 | 25 (24) | 14 (18)
  12 | 27 (23) | 22 (24)
  24 | 28 (22) | 13 (18)
  36 | 36 (22) | 15 (19)
  48 | 23 (19) | 12 (17)
Statistical Analysis 1: Comparison: Cesarean Delivery vs Vaginal Delivery; Pain at rest 6 h; Test type: Other; p = 0.06, Kruskal-Wallis
Statistical Analysis 2: Comparison: Cesarean Delivery vs Vaginal Delivery; Pain at rest 12 h; Test type: Other; p = .30, Kruskal-Wallis
Statistical Analysis 3: Comparison: Cesarean Delivery vs Vaginal Delivery; Pain at rest 24 h; Test type: Other; p = .002, Kruskal-Wallis
Statistical Analysis 4: Comparison: Cesarean Delivery vs Vaginal Delivery; Pain at rest 36 h; Test type: Other; p = 0.003, Kruskal-Wallis
Statistical Analysis 5: Comparison: Cesarean Delivery vs Vaginal Delivery; Pain at rest at 48 h; Test type: Other; p = .02, Kruskal-Wallis

3. Secondary Outcome: Satisfaction Scores
Description: This outcome will be measured using a visual analogue score (VAS). Patient will mark their satisfaction on a 0-100 mm line with 0 been not satisfied at all and 100 mm extremely satisfied.
Time Frame: 6 hours following delivery until 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Cesarean Delivery | Vaginal Delivery
Number analyzed (Participants) | 25 | 25
score on a scale (0-100)
  6 | 71 (34) | 78 (31)
  12 | 69 (29) | 80 (28)
  24 | 60 (32) | 83 (30)
  36 | 58 (29) | 95 (13)
  48 | 57 (32) | 89 (27)
Statistical Analysis 1: Comparison: Cesarean Delivery vs Vaginal Delivery; Satisfaction with pain control 6 h; Test type: Other; p = .43, Kruskal-Wallis
Statistical Analysis 2: Comparison: Cesarean Delivery vs Vaginal Delivery; Satisfaction with pain control 12 h; Test type: Other; p = .24, Kruskal-Wallis
Statistical Analysis 3: Comparison: Cesarean Delivery vs Vaginal Delivery; Satisfaction with pain control 24 h; Test type: Other; p = .012, Kruskal-Wallis
Statistical Analysis 4: Comparison: Cesarean Delivery vs Vaginal Delivery; Satisfaction with pain control 36 h; Test type: Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 5: Comparison: Cesarean Delivery vs Vaginal Delivery; Satisfaction with pain control 48 h; Test type: Other; p = .0005, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Normal Spontaneous Vaginal Delivery | Cesarean Delivery
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
Small sample size. No standardized post-delivery ambulation protocol at any of the institutions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02967016/Prot_SAP_000.pdf